CLINICAL TRIAL: NCT05268315
Title: Acceptability and Feasibility of a Brief Psychoeducational Intervention for Parents of Children With Childhood Cancer
Brief Title: A Brief Parental Intervention on Learning and Education in Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Hyundai Hope On Wheels (Other)
Responsible Party: Principal Investigator, Eric Zimak, Clinical Assistant Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-224
Record Dates: First submitted 2022-02-02; First posted 2022-03-07 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Psychoeducational Intervention (Experimental): Parents of children with cancer who complete the study participate in a brief, 1-session psychoeducational intervention.
  Interventions: Behavioral: Brief Psychoeducational Intervention

INTERVENTIONS:
Behavioral: Brief Psychoeducational Intervention — The 1-session psychoeducational intervention is divided into three brief modules. Topics that are covered include thinking, learning, emotional, and behavioral functioning as they relate to childhood cancer, educational and school supports, and the role of neuropsychological and school-based assessments.

SUMMARY:
The purpose of this study is to assess whether a brief intervention about learning and education is both practical and acceptable for parents of children with cancer.

DETAILED DESCRIPTION:
After being provided details about the study, participants signing the study consent form complete pre-intervention questionnaires. Participants then complete a brief psychoeducational intervention, via a HIPAA-compliant web and video conferencing platform on Zoom. The intervention is followed by completion of a post-intervention evaluation form. The consent form and study questionnaires are completed through Research Electronic Data Capture (REDCap), a secure web-based application.

ELIGIBILITY:
Inclusion Criteria:

* parent(s) or legal guardian(s) of children with cancer
* preferred language for oral and written communication is English
* 18 years of age or older
* 1 or 2 parents or legal guardians can participate for each child

The child must also meet the following for the parent(s)/legal guardian(s) to participate:

* diagnosis of cancer
* child is actively receiving cancer treatment at University of New Mexico Hospital or recently completed treatment (within 0-6 months post-treatment)
* child is between the age of 3 and 14
* child resides in New Mexico

Exclusion Criteria: Parents of children who are wards of the state are excluded (including children in custody of the NM Children, Youth & Families Department).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of study recruitment and enrollment | Through study completion, up to 2 years
  Among qualifying families, the number receiving recruitment information about the study, identifying interest, scheduling, and completing procedures. Note, for each qualifying family, one or two parents or legal guardians are able to enroll in the study. This is a parental intervention and the child with cancer does not participate in the study.
Fidelity to the intervention protocol | at time of intervention (day 1)
  Interventions are audio-recorded. Percent adherence to the intervention protocol per a fidelity form, developed for this study, is assessed by an independent rater of fidelity.
Acceptability of the intervention | immediately post-intervention (day 1)
  Ratings are provided on intervention acceptability as part of the Program Evaluation Form, a questionnaire developed for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Zimak, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

DOCUMENTS (1):
  • Informed Consent Form (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT05268315/ICF_000.pdf